CLINICAL TRIAL: NCT06491472
Title: Efficacy and Safety of Ivonescimab(AK112/SMT112) in Combination With Stereotactic Body Radiation Therapy and Chemotherapy in Patients With Pancreatic Cancer：A Single-arm, Open-label, Phase II Clinical Study
Brief Title: Ivonescimab(AK112/SMT112) in Combination With Stereotactic Body Radiation Therapy and Chemotherapy in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Akesobio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-004
Record Dates: First submitted 2024-06-27; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
Keywords: locally advanced or metastatic pancreatic cancer; Ivonescimab(AK112/SMT112); first-Line therapy; chemotherapy; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ivonescimab(AK112/SMT112)+SBRT+gemcitabine+nab-paclitaxel (Experimental): Ivonescimab(AK112/SMT112) (20mg/kg,Q3W) +gemcitabine(1000 mg/m²,IV, d1/8, Q3W)+nab-paclitaxel(25mg/m2, IV, d1/8, Q3W)
  +SBRT(5Gy *5 F)
  Interventions: Drug: Ivonescimab; Drug: Gemcitabine; Drug: Nab paclitaxel; Radiation: SBRT

INTERVENTIONS:
Drug: Ivonescimab — 20mg/kg,IV,d1,Q3W
  Other Names: AK112/SMT112
Drug: Gemcitabine — 1000mg/m2, IV, d1/8, Q3W
Drug: Nab paclitaxel — 125mg/m2, IV, d1/8, Q3W
Radiation: SBRT — 5Gy *5 F

SUMMARY:
This study is an open-label, single-arm Phase II clinical study to evaluate the efficacy and safety of ivonescimab(AK112/SMT112) in combination with stereotactic body radiation therapy and chemotherapy in patients with pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent and comply with all requirements of study participation (including all study procedures).
* Histologically- or cytologically-confirmed diagnosis of pancreatic ductal adenocarcinoma (including adenosquamous carcinoma)
* Have a life expectancy of at least 3 months.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by investigator
* No previous history of radiotherapy or no overlap between the secondary radiotherapy site and the original radiotherapy site
* Has adequate organ function
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Has known active brain metastases or meningeal metastases
* Compression fractures of the spine not treated with surgery and/or radiation; Treated spinal compression fractures require stable disease for at least 2 weeks randomization
* There was a high risk of gastrointestinal bleeding or abdominal bleeding
* Uncontrolled cancer pain; Anesthetic painkillers did not reach a stable dose at the time of enrollment
* During the initial 72 hours of the study, patients experienced a weight loss of 10 percent or more compared to their initial body weight when they signed the ICF
* Within 72 hours prior to the study, the subjects' ECOG physical status score increased by ≥1 point compared to the score at ICF signing.
* Unable to lie flat or for 10-20 minutes with radiotherapy.
* Prior exposure to any agent targeting T cell costimulation or immune checkpoint pathways (e.g., anti-PD 1, anti-PD L1, anti-PD L2, anti-CTLA 4, anti CD137 or anti-OX40 antibody, etc)
* Known germ line BRAC1/2 mutation
* Liver metastases account for more than 50% of the total liver volume
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years before the first dose of study treatment;
* Received chemotherapy, tyrosine kinase inhibitors, immunotherapy (such as interleukin, interferon or thymosin) and other anti-tumor therapy within 28 days before the study, and received Chinese medicine with anti-tumor indications within 14 days before the administration
* Has undergone major surgery within 30 days prior to the first dose of study treatment
* Has received radical radiotherapy within 3 months before the study; Palliative radiotherapy was allowed 2 weeks before administration, and the radiotherapy dose was in line with local palliative treatment standards
* Systemic corticosteroids (>10 mg/ day of prednisone or equivalent equivalent of other corticosteroids, continuous treatment ≥7 days) or immunosuppressant therapy were required during the first 14 days of the study; Except inhaled or topical use of hormones, or physiological replacement dose of hormone therapy due to adrenal insufficiency; Short-term (≤7 days) corticosteroids are permitted for prevention (e.g., contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity caused by exposure to allergens)
* has a decline in albumin that was difficult to correct
* Has received a live virus vaccine within 28 days prior to first dose of study treatment.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Has an active infection requiring systemic therapy
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 6 months prior to day 1 of study treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator
* Has received a live virus vaccine within 28 days prior to first dose of study treatment
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment.
* Other cases deemed inappropriate by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of first dosing till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall Survival(OS) | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1
Adverse event (AE) | Up to approximately 2 years
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results
Duration of Response(DOR) | Up to approximately 2 years
  Time from first documented response (CR or PR) until documented disease progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital of China, Wuhan, China